CLINICAL TRIAL: NCT03896321
Title: Coronary Artery Ectasia in Elective Coronary Angiography : Predictors, Outcomes and Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Gamil Fathi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Coronary Artery Ectasia
Record Dates: First submitted 2019-03-23; First posted 2019-03-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Ectasia; Coronary Artery Disease
MeSH Terms: conditions — Dilatation, Pathologic; Coronary Artery Disease | interventions — Platelet Aggregation Inhibitors; Anticoagulants

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Asprin (Active Comparator): Patient will receive dual anti platelet asprin And clopidogrel
  Interventions: Drug: Antiplatelet Agents
- Clopidogrel (Active Comparator): Patient will receive dual anti platelet asprin And clopidogrel
  Interventions: Drug: Antiplatelet Agents
- Warfarin (Active Comparator): Patient will receive oral anticoagulation
  Interventions: Drug: Anticoagulants
- Novel oral anticoagulant (Active Comparator): Patient will receive oral anticoagulation
  Interventions: Drug: Anticoagulants

INTERVENTIONS:
Drug: Antiplatelet Agents — effect of dual antiplatelet in management of coronary artery ectasia
  Arms: Asprin; Clopidogrel
Drug: Anticoagulants — effect of oral anticoagulants in management of coronary artery ectasia
  Arms: Novel oral anticoagulant; Warfarin

SUMMARY:
Coronary artery ectasia (CAE) is the diffuse dilatation of coronary artery. It is defined as a dilatation with a diameter of 1.5 times the adjacent normal coronary artery . Its prevalence ranges from 1.2%-4.9% with male to female ratio of 3:1 .

Coronary ectasia likely represents an exaggerated form of expansive vascular remodelling (i.e. excessive expansive remodelling) in response to atherosclerotic plaque growth .

CAE is more common in males. Hypertension is a risk Factor. Interestingly, patients with DM have low incidence of CAE. This may be due to down regulation of MMP with negative remodelling in response to atherosclerosis . Smoking appears to be more common in patients with CAE than in those with coronary artery disease (CAD).

The angiographic classification for CAE (described by Markis et al.) categorizes the severity based on the extent of coronary arterial involvement: Type 1: Diffuse ectasia of 2-3 arteries; Type 2: Diffuse ectasia in one artery and localized in another; Type 3: Diffuse single arterial ectasia; Type 4: Localized or segmental ectasia .

Stable angina is the most common presentation in patients with CAE . Patients with CAE without stenosis had positive results during treadmill exercise tests. ST-elevation myocardial infarction (MI) , non-ST elevation MI can occur from altered blood flow by distal embolization or occlusion of ectatic segment with thrombus.

Medical management for CAE is a controversial area as there is lack of evidence based medicine, especially the role of antiplatelet versus anticoagulant agents. Aspirin was suggested in all patients because of coexistence of CAE with obstructive coronary lesions in the great majority of patients and the observed incidence of myocardial infarction, even in patients with isolated coronary ectasia .The role of dual anti platelet therapy has not been evaluated in prospective randomized studies. Based on the significant flow disturbances within the ectatic segments, chronic anticoagulation with warfarin as main therapy was suggested

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected CAD who are referred for elective coronary angiography

Exclusion Criteria:

* Previous admission with an acute coronary event, previous PCI or CABG.
* History of bleeding tendency or those with high bleeding risk according to the HAS-BLED bleeding risk score

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of dual antiplatelet therapy vs oral anticoagulants in patients with CAE - occurance of major adverse cardiovascular events | 6 months
  Efficacy endpoints defined as the occurance of major adverse cardiovascular events (MACE)
safety of dual antiplatelet therapy vs oral anticoagulants in patients with CAE - occurance of major or minor bleeding | 6 months
  safety endpoints of occurance of major or minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Salwa R. Demitry, Professor, Study Director — Assiut University
Locations (1):
- Martina Gamil, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code